CLINICAL TRIAL: NCT00919880
Title: A Phase II Randomized Clinical Trial of Neo-adjuvant Weekly Paclitaxel With or Without Carboplatin in Early Breast Cancer
Brief Title: Comparison of Neo-adjuvant Weekly Paclitaxel With or Without Carboplatin in Early Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B04
Record Dates: First submitted 2009-06-04; First posted 2009-06-12 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — CP protocol; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental)
  Interventions: Drug: carboplatin+ paclitaxel; Drug: paclitaxel
- Active Comparator (Active Comparator)
  Interventions: Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin+ paclitaxel — carboplatin AUC 2mg/mL*min/week, 3 week cycle up to 4 cycles; paclitaxel 80mg/m2/week, 3 week cycle up to 4 cycles
  Other Names: A
  Arms: Experimental
Drug: paclitaxel — paclitaxel 80mg/m2/week, 3 week cycle up to 4 cycles
  Other Names: B

SUMMARY:
The purpose of this study is to determine whether neo-adjuvant weekly paclitaxel with carboplatin is better than paclitaxel alone in efficiency and safety in early breast cancer, and to explore whether ultrasound and magnetic resonance imaging can predict the efficiency of neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* female patients between 18 and 65 years old
* pathological diagnosed invasive breast cancer; medium and high risk primary breast cancer according to St. Gallen 2007
* able and willing to give consent to participate in the study

Exclusion Criteria:

* pregnant or lactating females
* previous treatment for breast cancer
* other tumor history
* instable complication (e.g., myocardial infarction within 6 months, arrhythmia, unstable diabetes, hypercalcemia) or uncontrolled infection
* allergy history to similar drugs
* concurrent disease or condition that would make the patient inappropriate for study participation
* resist to participate in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
significant effect rate (the proportion of G4 and G5, graded by Miller & Payne Method); null effect rate (the proportion of G1 and G2) | within the first 14 days (plus or minus 3 days) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tianfeng Wang, Doctor, Study Chair — Beijing Cancer Hospital Breast Center
Locations (1):
- Beijing Cancer Hospital Breast Center, Beijing, Beijing Municipality, China